CLINICAL TRIAL: NCT06925048
Title: A Multi-cohort, Phase II Study of SHR0302 Combined With PD-1/PD-L1 Inhibition for Treatment naïve or Acquired Resistant to Immunology NSCLC
Brief Title: SHR0302 Combined With PD-1/PD-L1 Inhibition for Treatment naïve or Acquired Resistant to Immunology NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chunxia Su (Other)
Responsible Party: Sponsor-Investigator, Chunxia Su, Dr, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024LY1179
Record Dates: First submitted 2025-03-30; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer; JAK Inhibitor; Immunology
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1- maintenance treatment (Experimental): PD-1 inhibitor in combination with JAK inhibitor in the maintenance treatment
  Interventions: Drug: PD-1 inhbitor+SHR0302
- Arm2-Second line after first-line immunotherapy resistance (Experimental): PD-L1 inhibitor in combination with JAK inhibitor in the second line
  Interventions: Drug: PD-L1 inhibitor+SHR0302

INTERVENTIONS:
Drug: PD-1 inhbitor+SHR0302 — PD-1 inhbitor+SHR0302 in the maintenance treatment
  Arms: Arm1- maintenance treatment
Drug: PD-L1 inhibitor+SHR0302 — PD-L1 inhibitor+SHR0302 in second line
  Arms: Arm2-Second line after first-line immunotherapy resistance

SUMMARY:
Recent studies showed that the dysregulated activation of the JAK/STAT pathway, which leads to the prolonged release of IFN-γ, is a significant contributor to the resistance to immune checkpoint inhibitors in cancer immunotherapy. Preclinical and clinical studies have demonstrated that the combination of JAK inhibitors with PD-1 immunotherapy can reverse or delay onset of immunotherapy resistance by modulating the JAK/STAT pathway in Hodgkin's lymphoma and non - small cell lung cancer (NSCLC). SHR0302, being a highly selective JAK1 inhibitor, has shown excellent clinical benefits by effectively inhibiting the JAK/STAT pathway, leading to its approval for the treatment of Ankylosing Spondylitis in China. Preclinical studies also show that the combination of SHR0302 and PD-L1 inhibitor has synergistic potentials for anti-tumor effect in resistant to-immune checkpoint blockade patients. Thus, we conducted a phase 2 clinical trial evaluating SHR0302 combined with PD1/PD-L1 inhibitors as treatment-naïve or acquired resistant to first-line checkpoint inhibitor resistant NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Inoperable or non-suitable for radical radiotherapy and chemotherapy IIIB/IIIC and Stage IV or metastatic non-small cell lung cancer (NSCLC)
2. Provide written informed consent for the trial.
3. Patients ≥ 18 years of age
4. Arm 1: treatment naive; Arm 2: acquired resistant to first-line PD-1/PD-L1 inhibition. Acquired resistance is defined as documented initial objective response (partial or complete response by RECIST or WHO) to therapy or significant and durable (> 6 months) clinical benefit (stable disease defined by RECIST or WHO).
5. Subject must have adequate tumor burden at a safely accessible site for biopsy.
6. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
7. ECOG performance status 0 or 1
8. Adequate organ function:

(1) White Blood Cell ≥3.0×109/L; Absolute neutrophil count (ANC) ≥ 1.5×10*9 /L; Platelets ≥ 100×10*9 /L; Hemoglobin ≥ 9g/dl; (2) Serum creatinine ≤1.5 X upper limit of normal or creatinine clearance ≥ 40 mL/min; (3) Serum total bilirubin ≤ 1.5 X ULN; AST and ALT ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases; 9. Subjects of reproductive potential must agree to use acceptable birth control methods

Exclusion Criteria:

1. Non-small cell cancer contains components of small cell lung cancer or neuroendocrine carcinoma.
2. Sensitizing mutations in Epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) or ROS1 proto-oncogene receptor tyrosine kinase (ROS1) translocations;
3. Arm 1: Currently participating in or has participated in a study of an investigational agent or anticipated use of an investigational device within 4 weeks of the first dose of study treatment.
4. Receiving Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects within 2 weeks before the first administration.
5. Having a history of allergic reaction to any component of the study drug.
6. Having active hemoptysis requiring clinical intervention, active diverticulitis, abdominal abscess, gastrointestinal obstruction, and peritoneal metastasis.
7. Having clinically uncontrollable pleural effusion/abdominal effusion (patients who do not need to drain the effusion or whose effusion does not increase significantly within 3 days after stopping drainage can be enrolled).
8. The tumor compressing surrounding vital organs (such as the esophagus) and accompanied by related symptoms, compressing the superior vena cava or invading the large vessels in the mediastinum, the heart, etc.
9. Severe comorbidities such as a history of severe lung or heart diseases, and having experienced any arterial thrombosis, embolism, or ischemia within 6 months before being selected for treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, etc.
10. Having a history of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism within 3 months before enrollment.
11. Interstitial pneumonia (ILD), drug-induced pneumonia, radiation pneumonia requiring steroid treatment, or symptomatic active pneumonia.
12. Receiving systemic corticosteroids (>10 mg/d prednisone equivalent drugs) or other systemic immunosuppressants within 2 weeks before enrollment. Local, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids are allowed.
13. A history of autoimmune diseases. Patients with autoimmune-related hypothyroidism who are receiving a stable dose of thyroid hormone replacement therapy are eligible to participate in this study. Patients with type 1 diabetes mellitus who are under control after receiving a stable insulin treatment regimen are eligible to participate in this study.
14. Active systemic infection, including tuberculosis (clinical diagnosis includes clinical history, physical examination, and imaging findings, as well as TB examinations according to local medical routines), hepatitis B (known to be positive for HBV surface antigen (HBsAg) and HBV DNA ≥1000 cps/ml or the lower limit of its reference value), hepatitis C, or human immunodeficiency virus (positive for HIV antibody).
15. Known presence of mental illness or drug abuse that may affect compliance with the requirements of the trial.
16. Recently receiving sufficient oral or non-oral anticoagulants or thrombolytics. Prophylactic use of anticoagulants is allowed.
17. Having a medical history, disease, treatment, or laboratory abnormal results that may interfere with the trial results or prevent the subject from participating in the study throughout the whole process, or the investigator deems that participating in the study is not in the best interest of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 18 months
  PFS is defined as days from initiation of study therapy to first documented disease progression, death due to any cause or last subject contact which documents progression-free status.

SECONDARY OUTCOMES:
Objective response rate | percentage of evaluable subjects who achieve a complete or partial clinical response at 12 weeks
Duration of Response | through study completion, an average of 18 months
  DOR is defined as the time from first documentation of partial or complete response to first documented disease progression.
Overall survival | through study completion, an average of 18 months
  OS is defined as days from initiation of study therapy to death due to any cause or last subject contact.

IPD SHARING:
Plan to Share IPD: Yes